CLINICAL TRIAL: NCT06097962
Title: Exploratory Study of NK510 Combined With PD-1 Blockade in the Treatment of Relapsed and Refractory Advanced NSCLC
Brief Title: Safety and Efficacy of NK510 to Treat NSCLC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: The General Hospital of Eastern Theater Command (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NK510-06
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: NSCLC
MeSH Terms: interventions — sugemalimab

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (low-dose group) (Experimental): NK510 will be administered once a week for a total of six weeks.1×10^9 NK cells/dose.
  PD-1 blockade will be administered every 3 weeks.
  Interventions: Drug: NK510; Drug: Tislelizumab，atezolizumab or sugemalimab
- Group B (medium-dose group) (Experimental): NK510 will be administered once a week for a total of six weeks.9×10^9 NK cells/dose.
  PD-1 blockade will be administered every 3 weeks.
  Interventions: Drug: NK510; Drug: Tislelizumab，atezolizumab or sugemalimab
- Group C (high-dose group) (Experimental): NK510 will be administered once a week for a total of six weeks.12×10^9 NK cells/dose.
  PD-1 blockade will be administered every 3 weeks.
  Interventions: Drug: NK510; Drug: Tislelizumab，atezolizumab or sugemalimab

INTERVENTIONS:
Drug: NK510 — Intravenous infusion
Drug: Tislelizumab，atezolizumab or sugemalimab — Administer according to the instructions

SUMMARY:
This study will evaluate the safety and efficacy of NK510 in the treatment of relapsed and refractory advanced NSCLC.NK510 will be administered in combination with PD-1 blockade. Patients are required to undergo a biopsy for confirmation of tumor PD-L1 expression,and EGFR,ROS1,ALK gene must be negative. The safety and efficacy of this treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years;
* Epidermal growth factor receptor (EGFR) gene mutation negative, ROS oncogene 1 (ROS1) negative, and anaplastic lymphoma kinase (ALK) negative, stage III or IV non-small cell lung cancer that cannot be operated on or treated with radiotherapy, locally advanced or relapsed or metastatic non-small cell lung cancer;
* Biopsy tissue or pathological sections can be obtained, and tumor PD-L1 expression is positive (defined as ≥ 1% of TPS);
* After receiving ≥ 4 courses of PD-1 monoclonal antibody ± chemotherapy in the past, the disease is currently in a stable or progressive state;
* According to RECIST v1.1 (Solid Tumor Efficacy Evaluation Criteria), there is at least one CT scan measurable lesion present;
* ECOG physical status score of 0-2;
* Expected survival >=3 months;
* Except for hair loss and fatigue, all AE after anti-tumor treatments have alleviated toxicity to level 1 (CTCAE v5.0) or original baseline;
* Female of childbearing age must be non lactating and have a negative serum pregnancy test within 1 week prior to enrollment;
* Voluntarily sign an informed consent form to participate in this study.

Exclusion Criteria:

* Pregnant or lactating female patients;
* Patients with central nervous system metastasis (CNS) and/or cancerous meningitis and obvious symptoms;
* Other malignancies have been diagnosed within 3 years prior to the first use of the study drug;
* Subjects with active, known or suspected autoimmune diseases [excluding type I diabetes, hypothyroidism requiring hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis or alopecia) or diseases that are not expected to recur without external triggers;
* subjects have a history of immune deficiency, including HIV testing positive, or other acquired or congenital immune deficiency diseases or organ transplantation history;
* Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, etc; At rest, the QTc interval obtained from a 12 lead electrocardiogram examination is>480 ms; Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months prior to enrollment; The New York Heart Association (NYHA) has a heart function rating of ≥ II or a left ventricular ejection fraction (LVEF) of<50%; Clinically uncontrollable hypertension;
* Radical radiotherapy was performed within 4 weeks prior to enrollment; Local palliative radiotherapy or Chinese herbal medicine/traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before enrollment;
* Not fully recovered from major surgery or trauma within 2 weeks prior to enrollment;
* Participated in research drug trials and received research treatment or used research instruments within 4 weeks before enrollment;
* Other anti-tumor treatments outside of this research protocol are currently underway or planned;
* Received blood transfusion, erythropoietin, granulocyte colony stimulating factor (G-CSF), or granulocyte macrophage colony stimulating factor treatment within 2 weeks prior to enrollment;
* Subjects who received systemic treatment with corticosteroids (prednisone>10 mg/day or equivalent) or other immunosuppressive/enhancing drugs (such as thymosin, interleukin-2, and interferon) within 2 weeks prior to enrollment. Allowing selected subjects to inhale or topically use corticosteroids in the absence of active autoimmune diseases;
* The virological examination of hepatitis B or hepatitis C during screening meets any of the following criteria:

  1. HBsAg positive and peripheral blood HBV-DNA titer detection≥1×10^3 copies/mL or upper limit of normal value;
  2. HCV antibody positive;
* Subjects who are known to be allergic or intolerant to PD-1 monoclonal antibody.
* Meet any of the following standards:

  1. Hematological:Neutrophil count <1.5×10^9/L; Platelet count < 75×10^9/L; Hemoglobin < 9 g/dL;
  2. Hepatic:ALT > 3 × ULN (tumor liver metastasis ≥ 5×ULN); AST > 3×ULN (tumor liver metastasis ≥ 5×ULN); TBIL > 1.5 ×ULN or TBIL>2.5 × ULN (3.0 mg/dL) in Gilbert syndrome subjects;
  3. Renal:Serum creatinine > 1.5 × ULN or creatinine clearance < 50mL/min;
* Any uncertain factors that affect the safety or compliance of patients.
* Investigators believe that any other serious or uncontrollable medical disease, active infection, abnormal physical examination, laboratory examination, mental state change, or mental illness increases the risk of the subject or affects the research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | 6 weeks
  To evaluate the DLT during N510 treatment
Maximal Tolerable Dose | 6 weeks
  to evaluate the MTD of NK510

SECONDARY OUTCOMES:
Overall response rate (ORR) after administration | 6 weeks
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Tangfeng Lv, PhD, Principal Investigator — The General Hospital of Eastern Theater Command
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No